CLINICAL TRIAL: NCT06159998
Title: New Markers for Treatment Response to Radiotherapy in Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Study closed
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Cyrill Rentsch, MD-PhD, University of Basel
Other Study IDs: EKBB 180/09; 180/09 (Other: EKBB)
Record Dates: First submitted 2012-12-11; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: radiotherapy; markers
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * PBMCs
  * Sera
  * Urine
  * prostate cells in urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The actual follow-up of patients undergoing definite radiotherapy for prostate cancer includes regular measurements of prostate specific antigen (PSA). Successful radiotherapy is critically dependent on local control of cancer; however, PSA takes 2-3 years to reach a nadir after therapy. We aim at collecting blood/urine after prostate massage before, and after radiotherapy in order to define new markers predicting local control earlier and more precisely than PSA.

DETAILED DESCRIPTION:
Patients will be closely followed for 5 years (weeks 0, 2, 4, 6, and months 2, 3, 6, 9, 12, 18, 24, and then yearly). Each assessment includes PSA measurement, urine collection after prostatic massage, and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing radiotherapy of biopsy confirmed clinically localised adenocarcinoma of the prostate

Exclusion Criteria:

* patients with inflammatory processes of the rectum
* patients with no rectum due to previous surgery

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men undergoing definite radiotherapy for prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Bio-repository | first assessment using predifined markers after recruitment of 15 patients followed for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cyrill A Rentsch, MD-PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Urology, University Hospital Basel, Basel, Canton of Basel-City, Switzerland